CLINICAL TRIAL: NCT04407507
Title: Multicenter, Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy, Safety and Tolerability of Ivermectin in Mild Virus-positive Subjects (SARS-CoV)-2 With or Without Symptoms
Brief Title: Efficacy, Safety and Tolerability of Ivermectin in Subjects Infected With SARS-CoV-2 With or Without Symptoms
Acronym: SILVERBULLET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SARS-COV-IverMX-01
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
Keywords: Ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivermectin (Experimental): Ivermectin 12 mg / day for 3 days, in combination with paracetamol therapy (500 mg QID) for 14 days
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): Ivermectin placebo 12 mg / day for 3 days, in combination with paracetamol therapy (500 mg QID) for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — ivermectin 12 mg / day for 3 days, in combination with standard paracetamol therapy (500 mg QID) for 14 days
  Arms: Ivermectin
Drug: Placebo — Placebo of ivermectin 12 mg / day for 3 days, in combination with standard paracetamol therapy (500 mg QID) for 14 days
  Arms: Placebo

SUMMARY:
This study aims to evaluate the efficacy, safety and tolerability of Ivermectin in patients with mild SARS-CoV-2 infection, in the rate of progression to severe 2019 novel coronavirus disease (COVID-19).

The primary efficacy endpoint is the proportion of participants with a disease control status defined as no progression of severe disease Hypothesis (H0): There is no difference between group A (ivermectin + paracetamol) and group B (ivermectin + paracetamol) in terms of the primary endpoint on day 14.

DETAILED DESCRIPTION:
In late 2019, an unidentified viral pneumonia was detected in Wuhan, China. Later, it was declared that it was pneumonia due to a new coronavirus. The World Health Organization (WHO) officially called it COVID-19 disease (Xie and Chen 2020).

Ivermectin is a broad-spectrum antiparasitic agent, developed to combat parasitic worms in veterinary use and in human medicine. This compound has been used orally in humans to treat filariasis, but is also effective against other worm-associated infections, as well as parasitic skin diseases and insect infections. It is approved for human use in several countries, to treat onchocerciasis, lymphatic filariasis, strongyloidiasis, and scabies, and recently in capillary pediculosis. When avermectins were discovered, they represented a new class of compounds that kill various ranges of disease-causing organisms, as well as pathogen vectors, inside and outside the body. Ivermectin is a semi-synthetic mixture of two chemically modified avermectins, comprising 80% 22,23-dihydroavermectin B1 and 20% 22,23-dihydroavermectin-B1b.

Other diseases that have been treated with ivermectin are: trichinosis, vector insects, malaria, trypanosomiasis, allergic asthma, rosacea, bedbugs, schistosomiasis, chagas disease, epilepsy, neurological diseases. Furthermore, it has been observed to have effects as an antibiotic and anticancer (Crump 2017).

In turn, Ivermectin has been described as a broad-spectrum antiviral, inhibiting nuclear import by its ability to inactivate host nuclear transport proteins, such as integrase and nonstructural protein 5 (NS5), limiting the ability to infect the western virus of the Nile in low concentrations (Yang et al. 2020), as well as inhibiting the replication of the yellow fever virus and other flaviviruses, such as dengue, and encephalitis, probably attacking the activity of nonstructural helicase 3 (Crump 2017).

Ivermectin, at a dose of 150-200 mcg / kg, is the first line of treatment for river blind disease (onchocerca volvulus), lymphatic filariasis, and strongyloidiasis(Crump 2017)..

French authorities approved ivermectin for humans in 1987. Shortly thereafter, Merck & Co Inc donated ivermectin for onchocerciasis control. Since then, more than two billion treatments have been distributed in Africa and Latin America for onchocerciasis and lymphatic filariasis (Chaccour et al. 2013; Smit et al. 2016).

In this context, ivermectin adverse events have been mild, transient and associated with the intensity of the infection. No significant association was found between ivermectin plasma levels and adverse events(Merck & Co 2009).

Wagstaff et al. published preliminary studies in in vitro cultures, where they observed that a 5000-fold reduction in the viral RNA content of cells infected with the SARS-CoV-2 virus, treated with a single dose of ivermectin (Caly et al. 2020).

Ivermectin therapy has not been tested in COVID-19 subjects and is therefore intended to be used as an adjuvant treatment; therefore, all study subjects will receive ivermectin or placebo in addition to therapy that their treating physician deems appropriate. Since ivermectin is in an early phase of clinical development, the use of base therapy will ensure that all subjects, including subjects who are randomized to receive placebo, have the benefit of receiving treatment with the base therapy that is available.

Research Objectives The main objective of this study is to evaluate the efficacy, safety and tolerability of ivermectin in patients with mild SARS-CoV-2 infection, in the rate of progression to severe COVID-19.

Secondary objectives

* Quantify the replication rate of the SARS-CoV-2 virus at days 5 and 14 after diagnosis quantitatively by real-time reverse transcription polymerase chain reaction (RT-PCR).
* Evaluate the presence and frequency of symptoms associated with COVID-19 disease (fever, cough, myalgia, fatigue, shortness of breath, headache, diarrhea, and expectoration) daily for 14 days.
* Investigate the presence of adverse events associated or not with the study drug for 14 days.
* Search for associations between the morbidities of the evaluated subjects and the intensity of the disease.
* Search for a relationship between medical history of bacille Calmette Guerin (BCG) vaccines and the intensity of the disease.
* Evaluate the frequency of death in the subjects, associated with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute severe respiratory syndrome due to SARS-CoV-12 coronavirus infection defined by RT-PCR.
* Asymptomatic, or with mild symptoms who are taking outpatient treatment of the disease.
* Signed Informed Consent.

Exclusion Criteria:

1. Patients with severe disease COVID-19.
2. Positive to proof of infection by some other virus such as influenza H1N1, SARS, etc.
3. Recurrent urinary tract infections.
4. Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST)> 5 times above its normal limits.
5. Pregnant or lactating patients
6. Patients receiving antihypertensive medication verapamil, the immunosuppressant cyclosporin A and / or the antipsychotic trifluoperazine.
7. Patients with a known allergy or hypersensitivity to dewormers.
8. Patients who are using an antioxidant supplement.
9. Patients with a history of filariasis, strongyloidiasis, scabies, river blindness, or any parasitic disease in the last twelve months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alma M Perez, MD, Principal Investigator — Centro de Investigación Farmacéutica Especializada de Occidente S.C.
Locations (1):
- Investigacion Biomédica para el Desarrollo de Fármacos S.A. de C.V., Zapopan, Jalisco, Mexico

REFERENCES:
- [Result] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Result] Chaccour CJ, Kobylinski KC, Bassat Q, Bousema T, Drakeley C, Alonso P, Foy BD. Ivermectin to reduce malaria transmission: a research agenda for a promising new tool for elimination. Malar J. 2013 May 7;12:153. doi: 10.1186/1475-2875-12-153. PMID 23647969
- [Result] Smit MR, Ochomo E, Aljayyoussi G, Kwambai T, Abong'o B, Bayoh N, Gimnig J, Samuels A, Desai M, Phillips-Howard PA, Kariuki S, Wang D, Ward S, Ter Kuile FO. Efficacy and Safety of High-Dose Ivermectin for Reducing Malaria Transmission (IVERMAL): Protocol for a Double-Blind, Randomized, Placebo-Controlled, Dose-Finding Trial in Western Kenya. JMIR Res Protoc. 2016 Nov 17;5(4):e213. doi: 10.2196/resprot.6617. PMID 27856406
- [Result] Xie M, Chen Q. Insight into 2019 novel coronavirus - An updated interim review and lessons from SARS-CoV and MERS-CoV. Int J Infect Dis. 2020 May;94:119-124. doi: 10.1016/j.ijid.2020.03.071. Epub 2020 Apr 1. PMID 32247050
- [Result] Yang SNY, Atkinson SC, Wang C, Lee A, Bogoyevitch MA, Borg NA, Jans DA. The broad spectrum antiviral ivermectin targets the host nuclear transport importin alpha/beta1 heterodimer. Antiviral Res. 2020 May;177:104760. doi: 10.1016/j.antiviral.2020.104760. Epub 2020 Mar 3. PMID 32135219
- [Derived] de la Rocha C, Cid-Lopez MA, Venegas-Lopez BI, Gomez-Mendez SC, Sanchez-Ortiz A, Perez-Rios AM, Llamas-Velazquez RA, Meza-Acuna AI, Vargas-Iniguez B, Rosales-Galvan D, Tavares-Valdez A, Luna-Gudino N, Hernandez-Puente CV, Milenkovic J, Iglesias-Palomares C, Mendez-Del Villar M, Gutierrez-Dieck GA, Valderrabano-Roldan CG, Mercado-Cerda J, Robles-Bojorquez JG, Mercado-Sesma AR. Ivermectin compared with placebo in the clinical course in Mexican patients with asymptomatic and mild COVID-19: a randomized clinical trial. BMC Infect Dis. 2022 Dec 8;22(1):917. doi: 10.1186/s12879-022-07890-6. PMID 36482326
- See also: Stromectol. FDA Approved Package Insert 2009 — http://www.accessdata.fda.gov/drugsatfda_docs/label/2009/050742s026lbl.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ivermectin | Placebo
Started | 33 | 33
Completed | 33 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin | Placebo | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 31 | 61
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.24 (14.48) | 36.82 (13.90) | 38.53 (14.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 7 | 11 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 19 | 19 | 38
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Mexico | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Disease Control Status Defined as no Disease Progression to Severe.
Description: The subject is considered to have progressed to severe illness when one or more of the following criteria are present:
  1. Breathing difficulty (≥30 breaths per minute);
  2. Resting oxygen saturation ≤93%;
  3. Severe complications such as: respiratory failure, need for mechanical ventilation, septic shock, non-respiratory organic failure.
Time Frame: 14 days
Population: Participants With a Disease Control Status Defined as no Disease Progression to Severe, 3 subjects of the Ivermectin arm group and 7 of the placebo were excluded of the efficacy analysis due to wrong criteria of inclusion (3 of ivermectin and 6 from placebo) and withdrawal of consent (1 in placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 30 | 26
Participants | 30 | 26

2. Secondary Outcome: SARS-CoV-2 Viral Load, at 5 and 14 Days
Description: To determine viral load indirectly, the Ct value of the SARS-COV-2 gene N was used on days 1, 5 and 14 of treatment, considering values greater than 37.5 as negative.
Time Frame: days 1, 5 and 14
Population: Only positive subjects are reported, since Ct is not reported in negative subjects, therefore there is no data available to analyze this criterion, as negative subjects are reported, the values for analysis decrease.
Measure: Mean (Standard Deviation); unit: Cycle threshold
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 30 | 26
Cycle threshold
  Day 1 | 26.17 (6.36) | 23.3 (5.15)
  Day 5: number analyzed (Participants) | 26 | 24
  Day 5 | 30.52 (4.21) | 28.5 (3.73)
  Day 14: number analyzed (Participants) | 21 | 20
  Day 14 | 33.74 (4.77) | 32.94 (4.74)

3. Secondary Outcome: Presence and Frequency of Symptoms Associated With the COVID-19 Disease
Description: Subjects were asked to answer a symptoms dairy during 14 days, where they recorded the presence of the following symptoms; fever, cough, muscular pain, fatigue, breath difficulty, headache, diarrhea, palpitations, expectoration and "Other", in the other question several subjects answer hypogeusia/ageusia, hyposmia/anosmia and backpain.
  The total of days anaylized were considered as 100%; 364 days for placebo patients(26 subjects x 14 days), and 420 for ivermectin subjects (30 subjects x 14 days), then the number of days reported correspond to de % of days when symptom was present.
Time Frame: 14 days
Population: Subjects were asked to answer a symptoms dairy during 14 days, where they recorded the presence of the following symptoms; fever, cough, muscular pain, fatigue, breath difficulty, headache, diarrhea, palpitations, expectoration and "Other", in the other question several subjects answer hypogeusia/ageusia, hyposmia/anosmia and backpain.
Measure: Number; unit: percentage of days
Arm/Group | Ivermectin | Placebo
Number analyzed (Participants) | 30 | 26
percentage of days
  Fever | 7.67 | 5.44
  Cough | 51.7 | 34.1
  Muscular pain | 29.5 | 24.6
  Fatigue | 45.4 | 38.1
  Breath difficulty | 16.7 | 14.9
  Headache | 32.3 | 26.9
  Palpitations | 13 | 9.74
  Expectoration | 25.7 | 17.5
  Diarrhea | 13 | 7.16
  Hypogeusia/ageusia | 18.9 | 8.31
  Hyposmia/anosmia | 19.4 | 10.9
  Backpain | 1.79 | 0.57
  Other | 28.6 | 14.3

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Ivermectin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/33
Other Adverse Events (participants affected / at risk) | 6/33 | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin (N=33) | Placebo (N=33)
HT Central nervous system and spinal cord infections (Nervous system disorders) | 1 (1) | 0 (0) — encephalitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin (N=33) | Placebo (N=33)
HLT RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
LLT Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
HLT Urinary tract infections (Renal and urinary disorders) | 2 (2) | 0 (0)
HLGT Epidermal and dermal diseases (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Maculo-papular pruritus
PF Vertigo (General disorders) | 1 (1) | 0 (0)
HLGT anxiety disorders and symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Anxiety
HLGT Inflammatory gastrointestinal diseases (Gastrointestinal disorders) | 1 (1) | 0 (0) — gastritis
LLT Otitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
LLT pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HLT Nasal congestion and inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Nasal congestion
LLT Hypertension (Vascular disorders) | 1 (1) | 1 (1)
HLGT Glucose metabolism disorders (including diabetes mellitus) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Hyperglycemia
SOC Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Leukocytosis
HLT Musculoskeletal pain and discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — low back pain
LLT acidity (Gastrointestinal disorders) | 0 (0) | 1 (1)
LLT elevated Lipase (Endocrine disorders) | 0 (0) | 1 (1)
LLT Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) — NAUSEA
SOC Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rash
PT Acid Peptic Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
LLT Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LLT Dizziness (General disorders) | 0 (0) | 1 (1)
LLT Tachycardia (Vascular disorders) | 0 (0) | 1 (1)
LLT Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT04407507/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT04407507/SAP_001.pdf